CLINICAL TRIAL: NCT03933020
Title: Impact of Physical Activity on Cognitive Outcomes in Youth With Pediatric-onset Multiple Sclerosis
Brief Title: Impact of Physical Activity on Cognitive Outcomes in Youth With Pediatric-Onset Multiple Sclerosis (POMS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient interest in participating (for adult patients), and lack of parental consent to participate (for pediatric patients)
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Microsoft Corporation (Industry)
Responsible Party: Principal Investigator, Rohini Samudralwar, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0247
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Pediatric Onset Multiple Sclerosis (POMS)
Keywords: Multiple Sclerosis; Cognitive Impairment; Physical activity
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Exercise Group (Experimental)
  Interventions: Device: VR active video game intervention; Behavioral: Educational session
- Control Group (Active Comparator)
  Interventions: Behavioral: Standard Management of Physical Activity

INTERVENTIONS:
Device: VR active video game intervention — The Microsoft VR active game program will consist of 3 weekly sessions of 45 minutes each combining 3 different types of exercise
  Arms: Exercise Group
Behavioral: Educational session — This consists of two education discussion sessions on the benefits of exercise for people with MS. The investigator MS specialists will conduct these sessions either by phone or at the time of a clinic visit and will also discuss difficulties encountered by participants with adherence.
  Arms: Exercise Group
Behavioral: Standard Management of Physical Activity — Routine discussion of lifestyle factors including physical activity during clinic visits
  Arms: Control Group

SUMMARY:
The purpose of this study is to to determine how implementing a home-based virtual reality video (VR) game exercise program in young people with Multiple Sclerosis(MS) can improve disability outcomes by measuring its impact on cognitive assessments (BICAMS), subjective measures of cognitive, physical and psychosocial disability, and motor assessments (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Pediatric-Onset MS (<18 years) according to the 2017 revised McDonald criteria (relapsing-remitting)
* Expanded Disability Status Scale (EDSS) ≤ 5.0
* Relapse free for the past 30 days (including no corticosteroids)
* No contraindications to physical activity, including pregnancy
* Participant and parent (if between 15 and 18 years of age) written informed consent.

Exclusion Criteria:

* History of visual provoked seizures
* EDSS > 5.0

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Garcia-Tarodo, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center,Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 2 enrolled participants were lost to follow up before they were assigned to an intervention; therefore, no participants "started" per the ClinicalTrials.gov definition of "started," which is "the number of participants assigned to each arm or group."
Groups:
- All Participants: The enrolled participants were lost to follow up before being assigned to any intervention.
Period: Overall Study
Arm/Group | All Participants
Started | 0
Received an Intervention | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected before the participants were assigned to an intervention, and the 2 enrolled participants were lost to follow up before they were assigned to an intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: After searching all records and contacting all team members, the age of one of the participants was not able to be determined.
  years
    number analyzed (Participants) | 1
    (all) | 19 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Brief International Cognitive Assessment for MS (BICAMS) - Symbol Digit Modalities Test (SDMT) [Mean (Standard Deviation); unit: score on a scale] — The Brief International Cognitive Assessment for MS (BICAMS) Symbol Digit Modalities Test (SDMT) is a measure of sustained attention, working memory, and information processing speed. It consists of single digits paired with abstract symbols. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 seconds. The score is reported as the number correct over the 90-second time span, and possible score ranges from 0 to 120, with a higher score indicating a better outcome.
  score on a scale | 61 (2.8)
Brief International Cognitive Assessment for MS (BICAMS) - California Verbal Learning test - II [Mean (Standard Deviation); unit: score on a scale] — The examiner reads a list of 16 words at a slightly slower rate than one item per second. Participants listen to the list and then report as many of the words as possible. After the first recall, the entire list is read again in the same order followed by a second attempt at recall. Altogether, there are five learning trials. The measure is reported as the total words recalled over trials 1 to 5. Total score ranges from 0 to 80, with a higher score indicating a better outcome.
  score on a scale | 61.5 (7.78)
Brief International Cognitive Assessment for MS (BICAMS) - Brief Visuospatial Memory Test (BVMT) [Mean (Standard Deviation); unit: score on a scale] — In this test, six abstract designs (in a 2 x 3 array) are presented for 10 seconds. The display is then removed from view and participants are required to draw the 2 x 3 array of figures from memory, with the correct shapes in the correct position. Each design receives from 0 to 2 points representing accuracy and location. There are three learning trials and the outcome measure is the total number of points earned over the three trials. Total score ranges from 0 to 36, with a higher score indicating a better outcome.
  score on a scale | 29 (4.2)
Anxiety and Depression and Indicated by Score on the Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: score on a scale] — Total score ranges from 0 to 42, with a higher score indicating greater anxiety and depression. Population: Data for this outcome measure were collected from only 1 participant.
  score on a scale
    number analyzed (Participants) | 1
    (all) | 11 (0)
Physical and psychological impact of MS as assessed by the Multiple Sclerosis Impact Scale-29 [Mean (Standard Deviation); unit: score on a scale] — Total score on the Multiple Sclerosis Impact Scale-29 (MSIS-29) ranges from 29-145, with a higher score indicating a greater impact of multiple sclerosis on day to day life. Population: Data for this outcome measure were only collected from 1 participant.
  score on a scale
    number analyzed (Participants) | 1
    (all) | 108 (0)
Fatigue as assessed by the Modified Fatigue Impact Scale (MFIS) [Mean (Standard Deviation); unit: score on a scale] — Total score on the MFIS ranges from 0 to 84, with a higher score indicating greater impact of fatigue on functioning. Population: Data for this outcome measure were collected for only 1 participant.
  score on a scale
    number analyzed (Participants) | 1
    (all) | 75 (0)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Symbol Digit Modalities Test (SDMT)
Description: A measure of sustained attention, working memory and information processing speed. The outcome measure is a numerical score.
Time Frame: 3 months
Population: Data for this outcome measure were not collected from any participant.
Groups:
- Exercise Group: Virtual reality (VR) active video game intervention: The Microsoft VR active game program will consist of 3 weekly sessions of 45 minutes each combining 3 different types of exercise
  Educational session: This consists of two education discussion sessions on the benefits of exercise for people with MS. The investigator MS specialists will conduct these sessions either by phone or at the time of a clinic visit and will also discuss difficulties encountered by participants with adherence.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Symbol Digit Modalities Test (SDMT)
Description: as for outcome 1
Time Frame: 6 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Symbol Digit Modalities Test (SDMT)
Description: as for outcome 1
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - California Verbal Learning Test - II (CVLT-II)
Description: A measure of verbal memory (immediate recall) including the first 5 recall trials. The outcome measure is a numerical score (.../80).
Time Frame: 3 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - California Verbal Learning Test - II (CVLT-II)
Description: as for outcome 4
Time Frame: 6 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - California Verbal Learning Test - II (CVLT-II)
Description: as for outcome 4
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Brief Visuospatial Memory Test (BVMT) - Revised
Description: A measure of visuo-spatial learning and delayed recall, using the first 3 recall trials. The outcome measure is a numerical total score (.../12).
Time Frame: 3 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Brief Visuospatial Memory Test (BVMT) - Revised
Description: as for outcome 7
Time Frame: 6 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Cognitive Disability as Assessed by the Brief International Cognitive Assessment for MS (BICAMS) - Brief Visuospatial Memory Test (BVMT) - Revised
Description: as for outcome 7
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Physical and Psychological Impact of MS as Assessed by the Multiple Sclerosis Impact Scale-29 (MSIS-29)
Description: 29-item self-report measuring the physical and psychological impact of MS from the patient's perspective during the previous 2 weeks. The assessment consists of 29 statements, each scored between 1 (not at all) and 5 (extremely), with a total score between 29 and 145.
Time Frame: 3 Month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Physical and Psychological Impact of MS as Assessed by the Multiple Sclerosis Impact Scale-29 (MSIS-29)
Description: as for outcome 10
Time Frame: 6 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Physical and Psychological Impact of MS as Assessed by the Multiple Sclerosis Impact Scale-29 (MSIS-29)
Description: as for outcome 10
Time Frame: 12 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Fatigue as Assessed by the Modified Fatigue Impact Scale (MFIS)
Description: 21-item self-report measuring the impact of fatigue on physical, cognitive and psychosocial aspects of MS during the previous 4 weeks. The assessment contains 21 statements, each scored between 0 (never) and 4 (almost always). Items can be aggregated into three subscales (physical, cognitive, and psychosocial) as well as into a total MFIS score. The physical subscale can range from 0 to 36. The cognitive subscale can range from 0 to 40. The psychosocial subscale can range from 0 to 8. The total MFIS score can range from 0 to 84.
Time Frame: 3 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Fatigue as Assessed by the Modified Fatigue Impact Scale (MFIS)
Description: as for outcome 13
Time Frame: 6 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Fatigue as Assessed by the Modified Fatigue Impact Scale (MFIS)
Description: as for outcome 13
Time Frame: 12 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Anxiety and Depression as Assessed by the Hospital Anxiety and Depression Scale (HADS)
Description: 14-item self-report measuring the degree of anxiety and depression in participants during the previous week. The assessment contains 14 statements, each scored between 3 (most of the time) and 0 (not at all). The score can be subdivided into a Depression scale that can range from 0 to 21, and an Anxiety scale, that can range from 0 to 21.
Time Frame: 3 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Anxiety and Depression as Assessed by the Hospital Anxiety and Depression Scale (HADS)
Description: as for outcome 16
Time Frame: 6 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Anxiety and Depression as Assessed by the Hospital Anxiety and Depression Scale (HADS)
Description: as for outcome 16
Time Frame: 12 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Distance Walked as Assessed by the Six Minute Walk Test (6MWT)
Description: the participant is instructed to walk for six minutes as quickly and safely as possible and the distance covered will be recorded
Time Frame: 6 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Distance Walked as Assessed by the Six Minute Walk Test (6MWT)
Description: as for outcome 19
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Number of Clinical Relapses
Description: Assessment at each clinic visit
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: New Activity on MRI (T2 Lesions, Gd+)
Description: Assessment at each MRI
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Safety of Implementing a VR Active Video Game Program at Home as Assessed by the Number of Self-reported Incidents That Occur During the Exercise Sessions, Including Falls or Physical Injuries.
Time Frame: 1 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Safety of Implementing a VR Active Video Game Program at Home as Assessed by the Number of Self-reported Incidents That Occur During the Exercise Sessions, Including Falls or Physical Injuries.
Time Frame: 3 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Safety of Implementing a VR Active Video Game Program at Home as Assessed by the Number of Self-reported Incidents That Occur During the Exercise Sessions, Including Falls or Physical Injuries.
Time Frame: 6 month
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Degree of Incorporation of Physical Activity Into Daily Life as Assessed by a Self Report Questionnaire
Time Frame: 6 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Degree of Incorporation of Physical Activity Into Daily Life as Assessed by a Self Report Questionnaire
Time Frame: 12 months
Population: Data for this outcome measure were not collected from any participant.
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: not collected
Description: Both participants were lost to follow up after the time of enrollment, before the intervention was assigned, and before any adverse events could be assessed; therefore, adverse were not monitored or assessed for this study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT03933020/Prot_SAP_000.pdf